CLINICAL TRIAL: NCT06385132
Title: GlobAl Psychological and Psychiatric prOfile in Glioblastoma and Head and Neck Cancer paTients
Brief Title: Psychological and Psychiatric prOfile in Glioblastoma and Head and Neck Cancer
Acronym: APPOINT
Status: Recruiting | Type: Observational
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Sponsor
Other Study IDs: 6447
Record Dates: First submitted 2024-04-05; First posted 2024-04-25 (Actual); Last update posted 2025-08-15 (Actual); Status verified 2025-08

CONDITIONS: Glioblastoma; Head and Neck Cancer
MeSH Terms: conditions — Glioblastoma; Head and Neck Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Psychological Tests' administration — to assess global psychological and psychiatric profile of patients affected by GBM and H&N-C by means of standardized questionnaires

SUMMARY:
Approximately 30% of cancer patients may experience psychopathological disorders. The most common psychopathological disorders in cancer patients are mood disorders, anxiety, depression, adjustment disorders, and suicidal ideation. Among depressive disorders, mixed depression, with the simultaneous presence of symptoms of both depressive and manic polarity, is associated to higher levels of chronicity, functional impairment and suicidality. These disorders can also be worsened by loneliness and demoralization.

Patients with head and neck cancer (H&N-C) and Glioblastoma multiforme (GBM) have high psychological and sometimes psychiatric comorbidity probably due to the severity, poor prognosis of these cancers and harsh treatment toxicities.

The most important protective factor for psychopathology is psychological resilience, which is "the capacity of a person to protect themselves and their mental health when facing life adversities," such as a GBM or H&N-C diagnosis. Resilience is influenced by the affective temperament, which refers to basic personality traits related to behavioral and emotional reactivity to environmental stimuli. It is believed to be biologically determined and relatively stable throughout life.

To date, the literature does not clarify the role of resilience and temperament in mediating the psychological profile of cancer patients. Furthermore, extensive profiling of the psychological and psychiatric profile of these patients at such a critical and pivotal moment in their journey is currently lacking in the literature.

Aim of this study is to evaluate global psychological and psychiatric profile of patients affected by GBM and H&N-C and the eventual fluctuation over time during RT course. Conducting an early and accurate screening for potential psychopathological issues will give the opportunity to avoid factors that could: worsen patient compliance, lead to suicidal risk, and increase hospitalizations.

The results obtained will be utilized for planning precocious psychological or psychiatric take-in-charge aimed at promoting psychological well-being of H&N-C and GBM patients.

ELIGIBILITY:
Inclusion Criteria:

* Consecutive glioblastoma and head and neck cancer patients undergoing a long course of radiotherapy
* Patients in adjuvant RT
* Patients in radiotherapy plus chemotherapy (RTCT) adjuvant regimen
* Ability to understand and complete the questionnaires
* Age > 18 years
* Informed consent signed

Exclusion Criteria:

* Age > 75 years
* Glioblastoma and head and neck cancer patients undergoing palliative radiotherapy
* Patients with inability to express informed consent
* Patients denying informed consent
* Patients affected by severe language deficits

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with histologically proven isocitrate dehydrogenase 1 wild-type (IDH-1wt) GBM, with either complete or incomplete resection, undergoing external beam radiotherapy with concurrent CT and treated by standard regimen will be enrolled in this study
  Patients with histologically proven H&NC, undergoing external beam radiotherapy with/without concurrent CT and treated by standard regimens will be enrolled in this study
Sampling Method: Probability Sample
Enrollment: 207 (Estimated)
Dates: Start 2024-05-02 (Actual); Primary Completion 2026-08-12 (Estimated); Study Completion 2026-10-31 (Estimated)

PRIMARY OUTCOMES:
Distress Thermometer | 18 months
  Distress Thermometer is a visual analogue tool rating personal distress during the past week on a scale from 0 (no distress) to 10 (extreme distress). Compared to psychological questionnaires, which are used as 'gold-standard' reference instruments (i.e., the Hospital Anxiety and Depression Scale), a DT cut-off score ≥ 4 identifies patients with emotional distress ('caseness').

SECONDARY OUTCOMES:
Brief Psychiatric Rating Scale | 18 months
  The Brief Psychiatric Rating Scale was developed to assess the severity of psychopathology symptoms. Administration times are brief, which makes it appropriate for use in clinical settings.
  Items are rated based on the clinician's or interviewer's observation of the patient's behavior, whereas the remaining symptoms are assessed using the information obtained during the interview. For the present protocol, the 24-item version will be used. Possible scores vary from 24 to 168, with lower scores indicating less severe psychopathology.

CONTACTS AND LOCATIONS:
Overall Officials: Loredana Dinapoli, Principal Investigator — Fondazione Policlinico Universitario A. Gemelli, IRCCS
Locations (1):
- Fondazione Policlinico Universitario A. Gemelli IRCCS, Roma, Italy